CLINICAL TRIAL: NCT02874495
Title: Anticipation Effect on Painful Phenomenons Linked to Rectal Distension for Patients With a Crohn's Disease in Remission: Functional MRI Study
Brief Title: Anticipation Effect on Painful Phenomenons Linked to Rectal Distension for Patients With a Crohn's Disease in Remission
Acronym: Douleur IRMf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC11.220
Record Dates: First submitted 2016-07-25; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Rectal Distension; Remission; Anticipation; Painful
MeSH Terms: conditions — Crohn Disease; Pain | interventions — Psychological Tests; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers: 22 persons.
  Interventions: Behavioral: Psychological tests; Device: Magnetic Resonance Imaging; Behavioral: Heart Rate Variability
- Patients with Crohn's disease: 22 patients.
  Interventions: Behavioral: Psychological tests; Device: Magnetic Resonance Imaging; Behavioral: Heart Rate Variability

INTERVENTIONS:
Behavioral: Psychological tests — Related to affective and cognitive dimensions of pain.
Device: Magnetic Resonance Imaging — With a certain or uncertain anticipation phase of distension (warning light) followed or not by a rectal distension at the pain threshold previously determined, and then a retrospective quotation of pain during distension and the fear of pain induced by anticipation. Structural MRI and rest of functional connectivity measure MRI.
  With measure of heart rate variability.
  Other Names: MRI
Behavioral: Heart Rate Variability — During MRI session, from the electrocardiographic signal. (measure of variations on R-R interval in milliseconds ms).
  Other Names: HRV

SUMMARY:
Crohn's disease goes along with an alteration of the quality of life, even in remission and has a negative impact on stress management linked to the pain and the health. Conversely, stress and psychological variables play a significant role in the pathogenesis of this disease. These interrelations reflects the link between the brain and the digestive tract, called brain-gut axis. The autonomic nervous system (ANS) is the neurological interface, relaying in a bidirectional way, informations between the digestive tract and the central nervous system (CNS).

Visceral information can thus modulate the functionnement of CNS's areas involved in pain management but also in the management of emotional and cognitive behaviours. Yet, numerous work demonstrate the existence of a dysfunction of the ANS during Crohn's disease, with a dysautonomia of the sympatho-vagal balance.

Human brain respond by advance before and during the application of a painful stimulus that enable the organism to regulate its nociceptive system in order to handle the aversive stimulus incoming, via the activation of brin areas managing the pain, or the raise of pain awareness.

The uncertain and not predictable nature of a painful crisis and/or an inflammatory relapse in a chronic disease like Crohn's disease can be the origin of an anticipating apprehension and anxiety, that could influence visceral perception (increasing it). Nevertheless, only few studies exists about the differential role of certain or uncertain anticipation of the pain, despite the fact that they are associated to different emotional, cognitive and behavioral responses, and the effect of anticipation on painful visceral perception, have not yet been studied for parents in remission of Crohn's disease.

The main goal is to search during certain and uncertain visceral anticipation, induced by distension of an intra-rectal balloon for persons suffering from Crohn's disease in remission, compared to control subjects, with an MRI functional study

ELIGIBILITY:
Inclusion Criteria:

* For patients :

  * Patients over 18 years and less than 60 years.
  * Right-handed.
  * Diagnosis of Crohn's disease established on clinical biological, endoscopic and anatomopathological criteria.
  * Ideal localization and/or diarrhea of Crohn's Disease, with an absence of rectal or anoperineal ravages past or presents in order to not do distension on rectal/ and anoperineal lesions.
  * Crohn's disease treatment authorize : 5-aminosalicylates since at least 4 weeks with a stable dose since at least 2 weeks ; immunosuppressive drugs since at least 12 weeks with a stable dose since at least 4 weeks ; anti-TNF since at least 3 months with a stable dose since at least 1 month ; absence of corticosteroid treatment since at least 15 days.
  * Clinical remission : Crohn's Disease Activity Index (CDAI) < 150 (Best 1976) and biological : normal CRP and faecal calprotectin < 100 g/g.
  * Patient able to understand and follow necessary commissions for the conduct of the clinical trial, and that have given his free written consent for this study.
  * Registered to a French social security.
  * The person won't be allow to participate simultaneously to another study and there won't be an exclusion period to participation to a clinical or therapeutic trial at the end of this study.
* For healthy volunteers

  * Patients over 18 years and less than 60 years.
  * Right-handed.
  * Paired with patients for sex and age.
  * Absence of digestive surgical or medical history except appendectomy, hysterectomy, cholecystectomy, inguinal hernia cure and/or femoral.
  * Absence of digestive symptomatology searched while a standardized interrogation.
  * Clinical digestive exam normal.
  * The person won't be allow to participate simultaneously to another study and there won't be an exclusion period to. participation to a clinical or therapeutic trial at the end of this study.
  * Registered to a French social security.
  * Registered to the national file of persons participating to biomedicals searches without direct individual profit.

Exclusion Criteria:

* Subjet under 18 years and more than 60 years.
* Counter-argument for MRI : presence of intra-corporeal ferro-magnetic particles, claustrophobia.
* Existence of a severe condition on general level (cardiac, respiratory, hematological, renal, hepatic, cancerous).
* Existence of an organic digestive affection (gastritis, gallstones, duodenal ulcer, megacolon, inflammatory colitis).
* Existence or history malignant gastrointestinal condition.
* History of abdominal digestive surgery except appendectomy, hysterectomy, cure of inguinal hernia)
* Recto-anal or périneal active pathology (haemorrhoid , anal fissure …).
* Presence of arectal fecal impaction.
* Patient included in an other clinical or therapeutic trial.
* Patient treated by a drug sensitive to modify sensitivity and/or digestive motor function.
* Patient regularly receiving psychotropic drugs (anxiolytics, sedatives, antidepressants, neuroleptics).
* Patient with a pathology that could modify visceral sensitivity like diabetes or neurodegenerative diseases.
* Persons concerned by articles L1121-5 to L1121-8 of CSP.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Crohn's disease
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | 30 minutes
  Activation of cortical cerebral structures involved in visceral pain and communication paths between them With a certain or uncertain anticipation phase of distension (warning light) followed or not by a rectal distension at the pain threshold previously determined, and then a retrospective quotation of pain during distension and the fear of pain induced by anticipation. Structural MRI and rest of functional connectivity measure MRI.
  With measure of heart rate variability.
Heart Rate Variability | 30 minutes
  During MRI session, from the electrocardiographic signal. (measure of variations on R-R interval in milliseconds ms).
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Questionnaire of personality inventory NEO-FFI (Bouvard, 2005)
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Questionnaire of depressive symptomatology CES-D (Center for Epidemiologic Studies-Depression Scale; Radloff, 1977)
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Anxiety inventory (STAI-Y of Spielberger)
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Pain Catastrophizing Scale of Sullivan 1995
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Pain Anxiety Symptoms Scale of Cracken 1992
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Fear of Pain Questionnaire of McNeil andRainwater ; 1998
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Visceral Sensitivity Index of Labus; 2004
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Questionnaire of Mindfulness, Walach 2006
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Questionnaire for uncertainty intolerance (Freeston 1994)
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  The Illness Attitude Scales, Dammen 1999
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Childhood Trauma Questionnaire of Bernstein 2003
Psychological tests | 45 minutes
  Related to affective and cognitive dimensions of pain :
  Ways of Coping Checklist Revised, adapted in French by Cousson 1996

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Bonaz, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Achard S, Salvador R, Whitcher B, Suckling J, Bullmore E. A resilient, low-frequency, small-world human brain functional network with highly connected association cortical hubs. J Neurosci. 2006 Jan 4;26(1):63-72. doi: 10.1523/JNEUROSCI.3874-05.2006. PMID 16399673
- [Background] Al-Chaer ED, Lawand NB, Westlund KN, Willis WD. Visceral nociceptive input into the ventral posterolateral nucleus of the thalamus: a new function for the dorsal column pathway. J Neurophysiol. 1996 Oct;76(4):2661-74. doi: 10.1152/jn.1996.76.4.2661. PMID 8899636
- [Background] Baciu MV, Bonaz BL, Papillon E, Bost RA, Le Bas JF, Fournet J, Segebarth CM. Central processing of rectal pain: a functional MR imaging study. AJNR Am J Neuroradiol. 1999 Nov-Dec;20(10):1920-4. PMID 10588119
- [Background] Baert F, Moortgat L, Van Assche G, Caenepeel P, Vergauwe P, De Vos M, Stokkers P, Hommes D, Rutgeerts P, Vermeire S, D'Haens G; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Mucosal healing predicts sustained clinical remission in patients with early-stage Crohn's disease. Gastroenterology. 2010 Feb;138(2):463-8; quiz e10-1. doi: 10.1053/j.gastro.2009.09.056. Epub 2009 Oct 8. PMID 19818785
- [Background] Benarroch EE. The central autonomic network: functional organization, dysfunction, and perspective. Mayo Clin Proc. 1993 Oct;68(10):988-1001. doi: 10.1016/s0025-6196(12)62272-1. PMID 8412366
- [Background] Berman SM, Naliboff BD, Suyenobu B, Labus JS, Stains J, Ohning G, Kilpatrick L, Bueller JA, Ruby K, Jarcho J, Mayer EA. Reduced brainstem inhibition during anticipated pelvic visceral pain correlates with enhanced brain response to the visceral stimulus in women with irritable bowel syndrome. J Neurosci. 2008 Jan 9;28(2):349-59. doi: 10.1523/JNEUROSCI.2500-07.2008. PMID 18184777
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701
- [Background] Biswal BB, Mennes M, Zuo XN, Gohel S, Kelly C, Smith SM, Beckmann CF, Adelstein JS, Buckner RL, Colcombe S, Dogonowski AM, Ernst M, Fair D, Hampson M, Hoptman MJ, Hyde JS, Kiviniemi VJ, Kotter R, Li SJ, Lin CP, Lowe MJ, Mackay C, Madden DJ, Madsen KH, Margulies DS, Mayberg HS, McMahon K, Monk CS, Mostofsky SH, Nagel BJ, Pekar JJ, Peltier SJ, Petersen SE, Riedl V, Rombouts SA, Rypma B, Schlaggar BL, Schmidt S, Seidler RD, Siegle GJ, Sorg C, Teng GJ, Veijola J, Villringer A, Walter M, Wang L, Weng XC, Whitfield-Gabrieli S, Williamson P, Windischberger C, Zang YF, Zhang HY, Castellanos FX, Milham MP. Toward discovery science of human brain function. Proc Natl Acad Sci U S A. 2010 Mar 9;107(10):4734-9. doi: 10.1073/pnas.0911855107. Epub 2010 Feb 22. PMID 20176931
- [Background] Bitton A, Dobkin PL, Edwardes MD, Sewitch MJ, Meddings JB, Rawal S, Cohen A, Vermeire S, Dufresne L, Franchimont D, Wild GE. Predicting relapse in Crohn's disease: a biopsychosocial model. Gut. 2008 Oct;57(10):1386-92. doi: 10.1136/gut.2007.134817. Epub 2008 Apr 7. PMID 18390994
- [Background] Blankstein U, Chen J, Diamant NE, Davis KD. Altered brain structure in irritable bowel syndrome: potential contributions of pre-existing and disease-driven factors. Gastroenterology. 2010 May;138(5):1783-9. doi: 10.1053/j.gastro.2009.12.043. Epub 2010 Jan 4. PMID 20045701
- [Background] Bonaz B, Plourde V, Tache Y. Abdominal surgery induces Fos immunoreactivity in the rat brain. J Comp Neurol. 1994 Nov 8;349(2):212-22. doi: 10.1002/cne.903490205. PMID 7860779
- [Background] Bonaz B, Tache Y. Induction of Fos immunoreactivity in the rat brain after cold-restraint induced gastric lesions and fecal excretion. Brain Res. 1994 Jul 25;652(1):56-64. doi: 10.1016/0006-8993(94)90316-6. PMID 7953723
- [Background] Bonaz B, Tache Y. Water-avoidance stress-induced c-fos expression in the rat brain and stimulation of fecal output: role of corticotropin-releasing factor. Brain Res. 1994 Mar 28;641(1):21-8. doi: 10.1016/0006-8993(94)91810-4. PMID 8019847
- [Background] Bonaz B, Riviere PJ, Sinniger V, Pascaud X, Junien JL, Fournet J, Feuerstein C. Fedotozine, a kappa-opioid agonist, prevents spinal and supra-spinal Fos expression induced by a noxious visceral stimulus in the rat. Neurogastroenterol Motil. 2000 Apr;12(2):135-47. doi: 10.1046/j.1365-2982.2000.00188.x. PMID 10771495
- [Background] Bonaz B, Baciu M, Papillon E, Bost R, Gueddah N, Le Bas JF, Fournet J, Segebarth C. Central processing of rectal pain in patients with irritable bowel syndrome: an fMRI study. Am J Gastroenterol. 2002 Mar;97(3):654-61. doi: 10.1111/j.1572-0241.2002.05545.x. PMID 11926209
- [Background] Bonaz B, Sabate JM. [Brain-gut axis dysfunction]. Gastroenterol Clin Biol. 2009 Feb;33 Suppl 1:S48-58. doi: 10.1016/S0399-8320(09)71525-8. French. PMID 19303539
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Bouin M, Plourde V, Boivin M, Riberdy M, Lupien F, Laganiere M, Verrier P, Poitras P. Rectal distention testing in patients with irritable bowel syndrome: sensitivity, specificity, and predictive values of pain sensory thresholds. Gastroenterology. 2002 Jun;122(7):1771-7. doi: 10.1053/gast.2002.33601. PMID 12055583
- [Background] Boureau F, Luu M, Doubrere JF, Gay C. [Construction of a questionnaire for the self-evaluation of pain using a list of qualifiers. Comparison with Melzack's McGill Pain Questionnaire]. Therapie. 1984 Mar-Apr;39(2):119-29. No abstract available. French. PMID 6729763
- [Background] Bouvard, M., Cottreaux, J. Protocoles et échelles d'évaluation en psychiatrie et en psychologie. 4ème Ed, 2005 Masson.
- [Background] Collins SM. Stress and the Gastrointestinal Tract IV. Modulation of intestinal inflammation by stress: basic mechanisms and clinical relevance. Am J Physiol Gastrointest Liver Physiol. 2001 Mar;280(3):G315-8. doi: 10.1152/ajpgi.2001.280.3.G315. PMID 11171612
- [Background] Cousson, F, Bruchon-Schweitzer, M, Quintard, B, Nuissier, J, Rascle N. Analyse multidimensionnelle d'une échelle de coping: validation française de la WCC (Ways of Coping Checklist). Psychologie Française 1996 ; 41: 155-164.
- [Background] Dammen T, Friis S, Ekeberg O. The Illness Attitude Scales in chest pain patients: a study of psychometric properties. J Psychosom Res. 1999 Apr;46(4):335-42. doi: 10.1016/s0022-3999(98)00127-5. PMID 10340232
- [Background] Ducrotté P, Bonaz B. Stress et tube digestif dans Stress, Pathologies et Immunité. Thurin JM et Bauman N. Ed Flammarion Médecine-Sciences, 2003 : p181-189.
- [Background] Fairhurst M, Wiech K, Dunckley P, Tracey I. Anticipatory brainstem activity predicts neural processing of pain in humans. Pain. 2007 Mar;128(1-2):101-10. doi: 10.1016/j.pain.2006.09.001. Epub 2006 Oct 27. PMID 17070996
- [Background] Faure C, Giguere L. Functional gastrointestinal disorders and visceral hypersensitivity in children and adolescents suffering from Crohn's disease. Inflamm Bowel Dis. 2008 Nov;14(11):1569-74. doi: 10.1002/ibd.20506. PMID 18521915
- [Background] Freeston, M. H., Rheaume, J., Letarte, H., Dugas, M. J., & Ladouceur, R. Why do people worry? Personality and Individual Differences, 1994, 17, 791-802.
- [Background] Geboes K, Collins S. Structural abnormalities of the nervous system in Crohn's disease and ulcerative colitis. Neurogastroenterol Motil. 1998 Jun;10(3):189-202. doi: 10.1046/j.1365-2982.1998.00102.x. No abstract available. PMID 9659662
- [Background] Gillanders S, Wild M, Deighan C, Gillanders D. Emotion regulation, affect, psychosocial functioning, and well-being in hemodialysis patients. Am J Kidney Dis. 2008 Apr;51(4):651-62. doi: 10.1053/j.ajkd.2007.12.023. PMID 18371541
- [Background] Graff LA, Walker JR, Clara I, Lix L, Miller N, Rogala L, Rawsthorne P, Bernstein CN. Stress coping, distress, and health perceptions in inflammatory bowel disease and community controls. Am J Gastroenterol. 2009 Dec;104(12):2959-69. doi: 10.1038/ajg.2009.529. Epub 2009 Sep 15. PMID 19755973
- [Background] Guthrie E, Jackson J, Shaffer J, Thompson D, Tomenson B, Creed F. Psychological disorder and severity of inflammatory bowel disease predict health-related quality of life in ulcerative colitis and Crohn's disease. Am J Gastroenterol. 2002 Aug;97(8):1994-9. doi: 10.1111/j.1572-0241.2002.05842.x. PMID 12190166
- [Background] Hagmann P, Jonasson L, Maeder P, Thiran JP, Wedeen VJ, Meuli R. Understanding diffusion MR imaging techniques: from scalar diffusion-weighted imaging to diffusion tensor imaging and beyond. Radiographics. 2006 Oct;26 Suppl 1:S205-23. doi: 10.1148/rg.26si065510. PMID 17050517
- [Background] Isaacs KL. How rapidly should remission be achieved? Dig Dis. 2010;28(3):548-55. doi: 10.1159/000320415. Epub 2010 Sep 30. PMID 20926885
- [Background] Kiebles JL, Doerfler B, Keefer L. Preliminary evidence supporting a framework of psychological adjustment to inflammatory bowel disease. Inflamm Bowel Dis. 2010 Oct;16(10):1685-95. doi: 10.1002/ibd.21215. PMID 20155849
- [Background] Labus JS, Mayer EA, Chang L, Bolus R, Naliboff BD. The central role of gastrointestinal-specific anxiety in irritable bowel syndrome: further validation of the visceral sensitivity index. Psychosom Med. 2007 Jan;69(1):89-98. doi: 10.1097/PSY.0b013e31802e2f24. PMID 17244851
- [Background] Lembo T, Munakata J, Mertz H, Niazi N, Kodner A, Nikas V, Mayer EA. Evidence for the hypersensitivity of lumbar splanchnic afferents in irritable bowel syndrome. Gastroenterology. 1994 Dec;107(6):1686-96. doi: 10.1016/0016-5085(94)90809-5. PMID 7958680
- [Background] Li J, Norgard B, Precht DH, Olsen J. Psychological stress and inflammatory bowel disease: a follow-up study in parents who lost a child in Denmark. Am J Gastroenterol. 2004 Jun;99(6):1129-33. doi: 10.1111/j.1572-0241.2004.04155.x. PMID 15180736
- [Background] Lix LM, Graff LA, Walker JR, Clara I, Rawsthorne P, Rogala L, Miller N, Ediger J, Pretorius T, Bernstein CN. Longitudinal study of quality of life and psychological functioning for active, fluctuating, and inactive disease patterns in inflammatory bowel disease. Inflamm Bowel Dis. 2008 Nov;14(11):1575-84. doi: 10.1002/ibd.20511. PMID 18512245
- [Background] Lomax AE, Fernandez E, Sharkey KA. Plasticity of the enteric nervous system during intestinal inflammation. Neurogastroenterol Motil. 2005 Feb;17(1):4-15. doi: 10.1111/j.1365-2982.2004.00607.x. PMID 15670258
- [Background] Mansfield P. Real-time echo-planar imaging by NMR. Br Med Bull. 1984 Apr;40(2):187-90. doi: 10.1093/oxfordjournals.bmb.a071970. No abstract available. PMID 6744006
- [Background] McCracken LM, Zayfert C, Gross RT. The Pain Anxiety Symptoms Scale: development and validation of a scale to measure fear of pain. Pain. 1992 Jul;50(1):67-73. doi: 10.1016/0304-3959(92)90113-P. PMID 1513605
- [Background] McNeil DW, Rainwater AJ 3rd. Development of the Fear of Pain Questionnaire--III. J Behav Med. 1998 Aug;21(4):389-410. doi: 10.1023/a:1018782831217. PMID 9789168
- [Background] Meregnani J, Clarencon D, Vivier M, Peinnequin A, Mouret C, Sinniger V, Picq C, Job A, Canini F, Jacquier-Sarlin M, Bonaz B. Anti-inflammatory effect of vagus nerve stimulation in a rat model of inflammatory bowel disease. Auton Neurosci. 2011 Feb 24;160(1-2):82-9. doi: 10.1016/j.autneu.2010.10.007. Epub 2010 Nov 11. PMID 21071287
- [Background] Mertz H, Naliboff B, Munakata J, Niazi N, Mayer EA. Altered rectal perception is a biological marker of patients with irritable bowel syndrome. Gastroenterology. 1995 Jul;109(1):40-52. doi: 10.1016/0016-5085(95)90267-8. PMID 7797041
- [Background] Minderhoud IM, Oldenburg B, Wismeijer JA, van Berge Henegouwen GP, Smout AJ. IBS-like symptoms in patients with inflammatory bowel disease in remission; relationships with quality of life and coping behavior. Dig Dis Sci. 2004 Mar;49(3):469-74. doi: 10.1023/b:ddas.0000020506.84248.f9. PMID 15139501
- [Background] Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med. 1990 Apr;14(1):68-78. doi: 10.1002/mrm.1910140108. PMID 2161986
- [Background] Ohlsson B, Sundkvist G, Lindgren S. Subclinical sympathetic neuropathy appears early in the course of Crohn's disease. BMC Gastroenterol. 2007 Aug 14;7:33. doi: 10.1186/1471-230X-7-33. PMID 17697346
- [Background] Pavlov VA, Wang H, Czura CJ, Friedman SG, Tracey KJ. The cholinergic anti-inflammatory pathway: a missing link in neuroimmunomodulation. Mol Med. 2003 May-Aug;9(5-8):125-34. PMID 14571320
- [Background] Pellissier S, Dantzer C, Canini F, Mathieu N, Bonaz B. Psychological adjustment and autonomic disturbances in inflammatory bowel diseases and irritable bowel syndrome. Psychoneuroendocrinology. 2010 Jun;35(5):653-62. doi: 10.1016/j.psyneuen.2009.10.004. Epub 2009 Nov 11. PMID 19910123
- [Background] Persoons P, Vermeire S, Demyttenaere K, Fischler B, Vandenberghe J, Van Oudenhove L, Pierik M, Hlavaty T, Van Assche G, Noman M, Rutgeerts P. The impact of major depressive disorder on the short- and long-term outcome of Crohn's disease treatment with infliximab. Aliment Pharmacol Ther. 2005 Jul 15;22(2):101-10. doi: 10.1111/j.1365-2036.2005.02535.x. PMID 16011668
- [Background] Petrak F, Hardt J, Clement T, Borner N, Egle UT, Hoffmann SO. Impaired health-related quality of life in inflammatory bowel diseases: psychosocial impact and coping styles in a national German sample. Scand J Gastroenterol. 2001 Apr;36(4):375-82. doi: 10.1080/003655201300051171. PMID 11336162
- [Background] Piche T, Ducrotte P, Sabate JM, Coffin B, Zerbib F, Dapoigny M, Hua M, Marine-Barjoan E, Dainese R, Hebuterne X. Impact of functional bowel symptoms on quality of life and fatigue in quiescent Crohn disease and irritable bowel syndrome. Neurogastroenterol Motil. 2010 Jun;22(6):626-e174. doi: 10.1111/j.1365-2982.2010.01502.x. Epub 2010 Apr 19. PMID 20403099
- [Background] Ploghaus A, Tracey I, Gati JS, Clare S, Menon RS, Matthews PM, Rawlins JN. Dissociating pain from its anticipation in the human brain. Science. 1999 Jun 18;284(5422):1979-81. doi: 10.1126/science.284.5422.1979. PMID 10373114
- [Background] Ploghaus A, Becerra L, Borras C, Borsook D. Neural circuitry underlying pain modulation: expectation, hypnosis, placebo. Trends Cogn Sci. 2003 May;7(5):197-200. doi: 10.1016/s1364-6613(03)00061-5. PMID 12757820
- [Background] Porro CA, Baraldi P, Pagnoni G, Serafini M, Facchin P, Maieron M, Nichelli P. Does anticipation of pain affect cortical nociceptive systems? J Neurosci. 2002 Apr 15;22(8):3206-14. doi: 10.1523/JNEUROSCI.22-08-03206.2002. PMID 11943821
- [Background] Posserud I, Syrous A, Lindstrom L, Tack J, Abrahamsson H, Simren M. Altered rectal perception in irritable bowel syndrome is associated with symptom severity. Gastroenterology. 2007 Oct;133(4):1113-23. doi: 10.1053/j.gastro.2007.07.024. Epub 2007 Jul 25. PMID 17919487
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Appl Psychol Meas 1977 ; 3 : 385-401.
- [Background] Reber SO, Obermeier F, Straub RH, Falk W, Neumann ID. Chronic intermittent psychosocial stress (social defeat/overcrowding) in mice increases the severity of an acute DSS-induced colitis and impairs regeneration. Endocrinology. 2006 Oct;147(10):4968-76. doi: 10.1210/en.2006-0347. Epub 2006 Jun 22. PMID 16794011
- [Background] Ritchie J. Pain from distension of the pelvic colon by inflating a balloon in the irritable colon syndrome. Gut. 1973 Feb;14(2):125-32. doi: 10.1136/gut.14.2.125. PMID 4696535
- [Background] Saper CB. The central autonomic nervous system: conscious visceral perception and autonomic pattern generation. Annu Rev Neurosci. 2002;25:433-69. doi: 10.1146/annurev.neuro.25.032502.111311. Epub 2002 Mar 25. PMID 12052916
- [Background] Schnitzler F, Fidder H, Ferrante M, Noman M, Arijs I, Van Assche G, Hoffman I, Van Steen K, Vermeire S, Rutgeerts P. Mucosal healing predicts long-term outcome of maintenance therapy with infliximab in Crohn's disease. Inflamm Bowel Dis. 2009 Sep;15(9):1295-301. doi: 10.1002/ibd.20927. PMID 19340881
- [Background] Schoepfer AM, Trummler M, Seeholzer P, Seibold-Schmid B, Seibold F. Discriminating IBD from IBS: comparison of the test performance of fecal markers, blood leukocytes, CRP, and IBD antibodies. Inflamm Bowel Dis. 2008 Jan;14(1):32-9. doi: 10.1002/ibd.20275. PMID 17924558
- [Background] Schweinhardt P, Bushnell MC. Pain imaging in health and disease--how far have we come? J Clin Invest. 2010 Nov;120(11):3788-97. doi: 10.1172/JCI43498. Epub 2010 Nov 1. PMID 21041961
- [Background] Seminowicz DA, Labus JS, Bueller JA, Tillisch K, Naliboff BD, Bushnell MC, Mayer EA. Regional gray matter density changes in brains of patients with irritable bowel syndrome. Gastroenterology. 2010 Jul;139(1):48-57.e2. doi: 10.1053/j.gastro.2010.03.049. Epub 2010 Mar 27. PMID 20347816
- [Background] Seminowicz DA, Mikulis DJ, Davis KD. Cognitive modulation of pain-related brain responses depends on behavioral strategy. Pain. 2004 Nov;112(1-2):48-58. doi: 10.1016/j.pain.2004.07.027. PMID 15494184
- [Background] Simren M, Axelsson J, Gillberg R, Abrahamsson H, Svedlund J, Bjornsson ES. Quality of life in inflammatory bowel disease in remission: the impact of IBS-like symptoms and associated psychological factors. Am J Gastroenterol. 2002 Feb;97(2):389-96. doi: 10.1111/j.1572-0241.2002.05475.x. PMID 11866278
- [Background] Sipponen T, Karkkainen P, Savilahti E, Kolho KL, Nuutinen H, Turunen U, Farkkila M. Correlation of faecal calprotectin and lactoferrin with an endoscopic score for Crohn's disease and histological findings. Aliment Pharmacol Ther. 2008 Nov 15;28(10):1221-9. doi: 10.1111/j.1365-2036.2008.03835.x. Epub 2008 Aug 26. PMID 18752630
- [Background] Song GH, Venkatraman V, Ho KY, Chee MW, Yeoh KG, Wilder-Smith CH. Cortical effects of anticipation and endogenous modulation of visceral pain assessed by functional brain MRI in irritable bowel syndrome patients and healthy controls. Pain. 2006 Dec 15;126(1-3):79-90. doi: 10.1016/j.pain.2006.06.017. Epub 2006 Jul 18. PMID 16846694
- [Background] Spaziani R, Bayati A, Redmond K, Bajaj H, Mazzadi S, Bienenstock J, Collins SM, Kamath MV. Vagal dysfunction in irritable bowel syndrome assessed by rectal distension and baroreceptor sensitivity. Neurogastroenterol Motil. 2008 Apr;20(4):336-42. doi: 10.1111/j.1365-2982.2007.01042.x. Epub 2007 Dec 19. PMID 18179607
- [Background] Spetalen S, Sandvik L, Blomhoff S, Jacobsen MB. Autonomic function at rest and in response to emotional and rectal stimuli in women with irritable bowel syndrome. Dig Dis Sci. 2008 Jun;53(6):1652-9. doi: 10.1007/s10620-007-0066-0. PMID 17990112
- [Background] Spielberger, C.D., Gorsuch, R., Lushene, R. 1983. The State-Trait Personality Inventory (STAI, Form Y), Palo Alto, CA, Consulting Psychologists Press.
- [Background] Sullivan, M.J.L., Bishop, S. and Pivik, J. The Pain Catastrophizing Scale: Development and validation. Psychol. Assess. 1995, 7: 524-532.
- [Background] Summerton CB, Longlands MG, Wiener K, Shreeve DR. Faecal calprotectin: a marker of inflammation throughout the intestinal tract. Eur J Gastroenterol Hepatol. 2002 Aug;14(8):841-5. doi: 10.1097/00042737-200208000-00005. PMID 12172403
- [Background] Talairach J and Tournoux P,
- [Background] Tang LY, Nabalamba A, Graff LA, Bernstein CN. A comparison of self-perceived health status in inflammatory bowel disease and irritable bowel syndrome patients from a Canadian national population survey. Can J Gastroenterol. 2008 May;22(5):475-83. doi: 10.1155/2008/109218. PMID 18478133
- [Background] Taylor CT, Keely SJ. The autonomic nervous system and inflammatory bowel disease. Auton Neurosci. 2007 Apr 30;133(1):104-14. doi: 10.1016/j.autneu.2006.11.005. Epub 2007 Jan 17. PMID 17234460
- [Background] Thompson SC. Will it hurt less if i can control it? A complex answer to a simple question. Psychol Bull. 1981 Jul;90(1):89-101. No abstract available. PMID 7267899
- [Background] Tibble J, Teahon K, Thjodleifsson B, Roseth A, Sigthorsson G, Bridger S, Foster R, Sherwood R, Fagerhol M, Bjarnason I. A simple method for assessing intestinal inflammation in Crohn's disease. Gut. 2000 Oct;47(4):506-13. doi: 10.1136/gut.47.4.506. PMID 10986210
- [Background] Tibble JA, Sigthorsson G, Bridger S, Fagerhol MK, Bjarnason I. Surrogate markers of intestinal inflammation are predictive of relapse in patients with inflammatory bowel disease. Gastroenterology. 2000 Jul;119(1):15-22. doi: 10.1053/gast.2000.8523. PMID 10889150
- [Background] van Orshoven NP, Andriesse GI, van Schelven LJ, Smout AJ, Akkermans LM, Oey PL. Subtle involvement of the parasympathetic nervous system in patients with irritable bowel syndrome. Clin Auton Res. 2006 Feb;16(1):33-9. doi: 10.1007/s10286-006-0307-x. PMID 16477493
- [Background] Van Oudenhove L, Vandenberghe J, Dupont P, Geeraerts B, Vos R, Dirix S, Bormans G, Vanderghinste D, Van Laere K, Demyttenaere K, Fischler B, Tack J. Abnormal regional brain activity during rest and (anticipated) gastric distension in functional dyspepsia and the role of anxiety: a H(2)(15)O-PET study. Am J Gastroenterol. 2010 Apr;105(4):913-24. doi: 10.1038/ajg.2010.39. Epub 2010 Feb 16. PMID 20160711
- [Background] Verma-Gandhu M, Bercik P, Motomura Y, Verdu EF, Khan WI, Blennerhassett PA, Wang L, El-Sharkawy RT, Collins SM. CD4+ T-cell modulation of visceral nociception in mice. Gastroenterology. 2006 May;130(6):1721-8. doi: 10.1053/j.gastro.2006.01.045. PMID 16697736
- [Background] Wagner M, Peterson CG, Ridefelt P, Sangfelt P, Carlson M. Fecal markers of inflammation used as surrogate markers for treatment outcome in relapsing inflammatory bowel disease. World J Gastroenterol. 2008 Sep 28;14(36):5584-9; discussion 5588. doi: 10.3748/wjg.14.5584. PMID 18810778
- [Background] Walach H., Buttenmuller, V., Kleinknecht N., Schmidt S. Measuring mindfulness - the Freiburg Mindfulness Inventory (FMI). Personnality and Individual Differences, 2006, 40:1543-1555.
- [Background] Weisenberg M, Schwarzwald J, Tepper I. The influence of warning signal timing and cognitive preparation on the aversiveness of cold-pressor pain. Pain. 1996 Feb;64(2):379-385. doi: 10.1016/0304-3959(95)00105-0. PMID 8740617